Validation of PET/MRI integrated system acquisition for cardiac applications

NCT02062008

Document Date: December 12, 2016

## Study Application (Version 1.5)

| 1.0 General Information | | |
|---|---|---|
| *Enter the full title of your study: | | |
| Validation of PET/MRI integrated system acquisition for cardiac applications | | |
| *Enter the study number or study alias | | |
| Validation of cardiac PET MR * This field allows you to enter an abbreviated version of the Study Title to quickly identify this study. | | |
| 2.0 Add Department(s) | | |
| 2.1 List the departments associated with this study. The Principal Investigator's departme should be Primary.: | nt | |
| Primary Department Name | | |
| UCSF - 147100 - M_Radiology | | |
| 3.0 List the key study personnel: (Note: external and affiliated collab<br>are not in the UCSF directory can be identified later in the Qualific | | |
| Key Study Personnel section at the end of the form) | 54110115 | f |
| Key Study Personnel section at the end of the form) 3.1 *Please add a Principal Investigator for the study: | | f |
| | | f |
| 3.1 *Please add a Principal Investigator for the study: | | <b>f</b> |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Resident | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Resident Fellow | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Resident Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. | | <b>f</b> |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Resident Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: A) Additional Investigators Acevedo-Bolton, Gabriel, PhD Other Investigator | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: A) Additional Investigators Acevedo-Bolton, Gabriel, PhD Other Investigator Bacharach, Stephen | | f |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: A) Additional Investigators Acevedo-Bolton, Gabriel, PhD Other Investigator | | |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: A) Additional Investigators Acevedo-Bolton, Gabriel, PhD Other Investigator Bacharach, Stephen Other Investigator Behr, Spencer C Other Investigator | | |
| 3.1 *Please add a Principal Investigator for the study: Hernandez Pampaloni, Jose Miguel MD, MD Select if applicable Department Chair Fellow If the Principal Investigator is a Fellow, the name of the Faculty Advisor must be supplied below. 3.2 If applicable, please select the Research Staff personnel: A) Additional Investigators Acevedo-Bolton, Gabriel, PhD Other Investigator Bacharach, Stephen Other Investigator Behr, Spencer C | | |

Dae, Michael W Other Investigator Gerstenfeld, Edward P M.D. Other Investigator Guccione, Julius M Ph.D. Other Investigator Haraldsson, Henrik Other Investigator Hernandez Pampaloni, Jose Miguel MD, MD Co-Principal Investigator Hope, Michael D Other Investigator Hope, Thomas A, MD Other Investigator Kanaya, Alka M Other Investigator Liu, Jing PhD Other Investigator Mukai, Kanae Other Investigator Mukai, Kanae Other Investigator Naeger, David M Other Investigator Ordovas, Karen G MD, MAS, MD Co-Principal Investigator Saloner, David A Ph.D., PhD Other Investigator Yeghiazarians, Yerem Other Investigator B) Research Support Staff Gao, Kenneth T Research Assistant Lorca, Maria Clara Research Assistant Tao, Dora H Research Assistant Verdin, Emily F Research Assistant Wong, Samantha A Research Assistant 3.3 \*Please add a Study Contact: Hernandez Pampaloni, Jose Miguel MD, MD Ordovas, Karen G MD, MAS, MD The Study Contact(s) will receive all important system notifications along with the Principal Investigator. (e.g. The project contact(s) are typically either the Study Coordinator or the Principal Investigator themselves). 3.4 If applicable, please add a Faculty Advisor/Mentor:

#### 3.5 If applicable, please select the Designated Department Approval(s):

Add the name of the individual authorized to approve and sign off on this protocol from your Department (e.g. the Department Chair or Dean).

### 4.0 Qualifications of Key Study Personnel

### 4.1 November, 2015 - NEW Definition of Key Study Personnel and CITI Training Requirements:

UCSF Key Study Personnel include the Principal Investigator, other investigators and research personnel who are directly involved in conducting research with study participants or who are directly involved in using study participants' identifiable private information during the course of the research. Key Personnel also include faculty mentors/advisors who provide direct oversight to Postdoctoral Fellows, Residents and Clinical Fellows serving as PI on the IRB application. The IRB requires that all Key Study Personnel complete Human Subjects Protection Training through CITI prior to approval of a new study, or a modification in which KSP are being added. More information on the CITI training requirement can be found on our website.

List the study responsibilities and qualifications of any individuals who qualify as Key Study Personnel (KSP) at UCSF and affiliated sites ONLY by clicking the "Add a new row" button. This information is required and your application will be considered incomplete without it.

| KSP Name | Description of Study<br>Responsibilities | Qualifications |
|---|---|---|
| Dr. Ordovas, Karen G MD, MD | Co-Principal Investigator, | Radiologist with large expertise in MRI cardiac applications |
| Dr. Saloner, David, PhD | Other Investigator, | PhD Physiscit. Expert in MRI applications in the cardiovascular system. |
| Lorca, Maria Clara | Research Assistant | Post- Doctoral Fellowship |
| Hernandez Pampaloni, Jose MD,<br>PhD, MD, PhD | Co-Principal Investigator | Radiologist. Chief of Nuclear Medicine at UCSF with extensive published work in cardiovasular PET imaging. |
| Behr, Spencer, MD | Other Investigator, | Radiologist with expertise in cross-sectional imaging |
| Botvinick, Elias H | Other Investigator, | Cardiologist. Expert in Nuclear<br>Cardiology |
| Liu, Jing PhD, PhD | Other Investigator, | PhD, Physicist. Expertise in cross-sectional physics |
| Dae, Michael W | Other Investigator, | Radiologist. Expert in nuclear cardiology |
| Acevedo-Bolton, Gabriel, PhD | Other Investigator, | PhD |
| Dr. Guccione, Julius, PhD | Other Investigator, | Bioengineer |
| Dr. Hope, Michael MD, MD | Other Investigator, | Chest Radiologist with |

| | | expertise in MRI applications in the cardiovascular field |
|---|---|---|
| Naeger, David M | Other Investigator, | Chest Radiologist. Expertise in PET imaging and cross-sectional imaging of the chest. |
| Dr. Yeghiazarians, Yerem MD,<br>1995 | Other investigator | Cardiologist. Interventional<br>Cardiologist |
| Dr. Kanaya, Alka MD | Other investigator | Cardiologist |
| Hope, Thomas A, MD | Other investigator | Radiologist with experience in PET and cross-sectional imaging |
| Dr. Gerstenfeld, Edward P M.D.<br>, MD | Other investigator | Cardiologist. Chief of cardiac electrophysiology |
| Dr. Haraldsson, Henrik PhD | Other investigator | Physicist |
| Bacharach, Stephen | Other Investigator | Physicist. Extensive experience in applications of PET imaging in cardiovascular disorders, including quantification of myocardial blood flow |
| Mukai, Kanae | Other investigator | Advanced Cardiac Imaging fellow |

#### Initial Screening Questions - Updated 9/13 5.0

(Note: You must answer every question on this page to proceed).

# 5.1 \* Application type: • Full Committee Expedited C Exempt 5.2 \* Risk level (Help Text updated 9/13): O Minimal risk Greater than minimal risk 5.3 \* Subject contact: • Yes (including phone, email or web contact) O No (limited to medical records review, biological specimen analysis, and/or data analysis) 5.4 \* Funding (past or present):

Funded or will be funded (external sponsor, gift, program or specific internal or departmental funds)

O Unfunded (no specific funds earmarked for this project)

| O Unfunded student project | |
|---|---|
| 5.5 * The Principal Investigator and/or one or more of the key study personnel has financial intercretated to this study: | ests |
| O Yes • No If <b>Yes</b> , the Conflict of Interest Advisory Committee (COIAC) office may contact you for additional information. | |
| 5.6 * This is an investigator-initiated study: | |
| ⊙ Yes O No | |
| 5.7 * This study ONLY involves retrospective records review and/or identifiable biospecimen analysis | ysis: |
| O Yes • No | |
| 5.8 * This is a clinical trial: | |
| 5.9 * This is a multicenter study: | |
| O Yes O No | |
| 5.10 * This application involves the study of unapproved or approved drugs, devices, biologics or i diagnostics: | in vitro |
| ⊙ Yes O No | |
| 5.11 * This application involves a Humanitarian Use Device: | |
| <ul><li>No</li><li>Yes, and it includes a research component</li><li>Yes, and it involves clinical careONLY</li></ul> | |
| 5.12 * This study involves human stem cells (including iPS cells and adult stem cells), gametes or embryos: | |
| <ul> <li>No</li> <li>Yes, and requires CHR and GESCR review</li> <li>Yes, and requires GESCR review, but NOT CHR review</li> </ul> | |
| 5.13 * This is a CIRB study (e.g. the NCI CIRB will be the IRB of record): | |
| O Yes O No | |

| No | | No is request is approved, the s of record. | e CHR will <b>NOT</b> review ar | nd approve t | his study. <i>i</i> | Another insti | tution will | |
|---|---|---|---|---|---|---|---|---|
| 6.0 | Fu | nding | | | | | | |
| 6.1 | only fund<br>docu | ify all sponsors and provine Prime Sponsor: ing coming through the Analysis of | Note: we require th UCSF. Please av Number if a P Nu d when a new fur ion or want these | only a P<br>void thes<br>umber wanding cyc<br>changes | Numbe<br>e comm<br>as alrea<br>le begir<br>made. | er <u>OR</u> an Androne<br>non errors<br>dy providus.<br>The IF | A Number s in fundin | for<br>g<br>date |
| Ex | ternal S | ponsor: | | | | | | |
| | View<br>Details | Sponsor Name | Sponsor Type | Awardee<br>Institution | Contract<br>Type: | UCSF RAS "P number" or eProposal number | UCSF<br>RAS<br>System<br>Award<br>Number<br>("A" +<br>6<br>digits) | |
| | Ξ | GE Medical Systems | 04 | UCSF | Grant | P0501481 | | |
| 3 | Sponsor | Name: | GE Medical Systems | | I | | | |
| | Sponsor | Type: | 04 | | | | | |
| 3 | Sponsor | Role: | Funding | Funding | | | | |
| | CFDA Nu | ımber: | | | | | | |
| | Grant/C | ontract Number: | CA-0050676 | | | | | |
| 1 | Awardee | Institution: | UCSF | | | | | |
| | ls Instit<br>Holder: | ution the Primary Grant | Yes | | | | | |
| ( | Contract | Type: | Grant | | | | | |
| | | S "P number" or<br>al number: | P0501481 | | | | | |
| | UCSF RAS System Award Number ("A" + 6 digits): | | | | | | | |
| | | umber for Studies Not<br>thru UCSF: | | | | | | |
| ( | Grant Ti | tle: | | | _ | | | |
| ( | PI Name<br>(If PI is on the st | not the same as identified | 1 | | | | | |
| 3 | Significa | nt Discrepancy: | | | | | | |

5.14 \* This application includes a request to rely on another IRB (other than NCI CIRB):

| Gift, Program, or Internal Funding (check all that apply): | |
|---|---|
| ☐ Funded by gift (specify source below) | |
| ☐ Funded by UCSF or UC-wide program (specify source below) | |
| lacksquare Specific departmental funding (specify source below, if applicable) | |
| List the gift, program, or departmental funding source: | |
| 6.2 If you tried to add a sponsor in the question above and it was not in the list, follow these step | s: |
| <ul> <li>6.2 If you tried to add a sponsor in the question above and it was not in the list, follow these steps:</li> <li>If funding has already been awarded or the contract is being processed by the Office of Sponsored Research (OSR) or Industry Contracts Division (ICD), your sponsor is already in the system and the project has an eProposal Proposal or Award number. Check with your department's OSR Staff or ICD Officer to ask how the sponsor is listed in the UC sponsor list and what the Proposal or Award number is. Click here to find your OSR staff and here to find your ICD staff.</li> <li>If your sponsor is not yet in the list, enter it in the box below.</li> </ul> | |
| C Sponsor not in list | |
| Only if your sponsor is not yet in the list, type the sponsor's name: | |
| If the funding is administered by the UCSF Office of Sponsored Research, your study will not receive CHR approval until the sponsor and funding details have been added to your application. | |
| 6.3 * This study is currently supported in whole or in part by Federal funding OR has received ANY Federal funding in the past (Help Text updated 9/13): | |
| O Yes • No | |
| If <b>yes</b> , indicate which portion of your grant you will be attaching: | |
| lacksquare The Research Plan, including the Human Subjects Section of your NIH grant or subcontract | |
| For other federal proposals (contracts or grants), the section of the proposal describing human subjects work | |
| ☐ The section of your progress report if it provides the most current information about your human subjects work | |
| ☐ The grant is not attached. The study is funded by an award that does not describe specific plans for human subjects, such as career development awards (K awards), cooperative agreements, program projects, and training grants (T32 awards) OR UCSF (or the affiliate institution) is not the prime recipient of the award | |
| 7.0 Sites | |
| 7.1 Institutions (check all that apply): | |
| ✓ UCSF | |
| ✓ China Basin | |
| Helen Diller Family Comprehensive Cancer Center | |
| ☐ Mission Bay | |
| Mount Zion | |
| ☐ San Francisco General Hospital (SFGH) ☐ SF VA Medical Center (SF VAMC) | |
| ☐ Blood Centers of the Pacific (BCP) | |

| ☐ Blood Systems Research Institute (BSRI) |
|---|
| Fresno (Community Medical Center) |
| ☐ Gallo ☐ Gladstone |
| ☐ Institute on Aging (IOA) |
| ☐ Jewish Home |
| SF Dept of Public Health (DPH) |
| 7.2 Check all the other types of sites not affiliated with UCSF with which you are cooperating or collaborating on this project (Help Text updated 9/13): |
| Other UC Campus |
| Other institution |
| ☐ Other community-based site |
| ☐ Foreign Country |
| List the foreign country/ies: |
| 7.3 Check any research programs this study is associated with: |
| ☐ Cancer Center |
| Center for AIDS Prevention Sciences (CAPS) |
| Global Health Sciences |
| ☐ Immune Tolerance Network (ITN) |
| <ul><li>□ Neurosciences Clinical Research Unit (NCRU)</li><li>□ Osher Center</li></ul> |
| Positive Health Program |
| 8.0 Study Design |
| 8.1 * Study design (Help Text updated 9/13): |
| The goal of this study is to understand how simultaneous PET/MR acquisition can provide novel qualitative and quantitative information to guide clinical intervention and predict prognosis of patients with risk factors for the development of coronary artery disease, or with diagnosis of cardiovascular ischemic or inflamatory disorders. |
| Patients required to have a clinical cardiac FDG PET or PET/CT imaging study as part of standard of care, to detect myocardial viability or a cardiac inflammatory process will be enrolled in the study. After the initial acquisition of the clinical study patients will be immediately imaged in the PET/MRI system, with no additional administration of any radiopharmaceutical. The main purpose of the study would then be to compare the infomration proveided form the clinical PET/CT with the one from the simultaneous cardiac PET/MRI. |
| 8.2 If this is a clinical trial, check the applicable phase(s) (Help Text updated 9/13): |
| □ Phase I □ Phase II □ Phase III □ Phase IV |
| 9.0 Scientific Considerations |

| 9.1 Hypothesis (Help Text updated 9/13): | |
|---|---|
| This study has a hypothesis: Yes O No If yes, state the hypothesis or hypotheses: We hypothesize that simultatenous acquisition of cardiac PET/MRI can could provide some other benefits in comparison to stand alone scanners. In a hybrid system, real-time MR-based motion detection and correction could be applied since cardiac and respiratory gating can be image-based without external sensors. This could allow partial-volume correction and event-based correction of patient motion during the PET acquisition. Combined metabolic information provided by FDG and structural information offered by MRI can help to better define the extent, location and significance of infarcted myocardium or viable tissue, with special significance for non-transmural or transmural lesions. The lack of exposure to ionizing radiation and iodinated contrast agents makes hybrid PET/MRI attractive when compared with PET/CT. Both cardiac MRI and PET examinations can be rather time consuming. Thus, improvements in patient compliance as a result of reduced scan time could be significant, particularly in patients with dyspnea due to heart failure who have difficulty holding their breath during MRI acquisitions. Increased patient throughout based on reduced scan times is also likely to be cost-effective. | |
| 9.2 * List the specific aims: | |
| <ul> <li>To compare regional myocardial uptake of FDG on images obtained on a standard PET camera with the new PET/MR camera, in patients with and without overt diagnosis of ischemic coronary artery disease.</li> <li>To compare viability maps obtained with cardiac MR images and FDG-PET for delineation of myocardial infarct core and border zone, in patients with coronary artery disease.</li> <li>To correlate MRI myocardial strain with relative myocardial FDG uptake in patients with a previous myocardial infarction, referred for a clinical myocardial viability study.</li> <li>To interrogate if simultaneous acquisition of cardiac PET and viability cardiac MR differ from acquisitions obtained independently, with special focus on attenuation correction methods.</li> <li>To combined MRI scar map with FDG-PET uptake in patients with cardiac sarcoidosis and myocarditis.</li> <li>To evaluate cardiac strain and myocardial scar burden in obese patients with and without diabetes.</li> </ul> | |
| 9.3 Statistical analysis: | |
| Correlation coefficient and Bland Altman plots will be applied to evaluate the agreement between linear variables obtained from PET and cardiac MRI. | |
| 9.4 If this study has undergone scientific or scholarly review, please indicate which entity performs review: | ed the |
| <ul> <li>□ Cancer Center Protocol Review Committee (PRC) (Full approval is required prior to final CHR approval for cancer-related protocols.)</li> <li>□ CTSI Clinical Research Center (CRC) advisory committee</li> <li>☑ Departmental scientific review</li> <li>□ Other:</li> <li>Specify Other:</li> </ul> | |

### 10.0 Background

#### 10.1 Background:

#### **Background**

Magnetic resonance (MR) imaging and positron emission tomography (PET) have been clinically available for more than 20 years and have evolved into highly valuable and versatile tools in diagnostic imaging. Since their first introduction, both imaging modalities have undergone a largely independent evolution in regard to technological development and clinical application. Nevertheless, since the first implementation of these inherently different imaging modalities, the idea of combining both into hybrid systems to complement each other has emerged.

Simultateous acquisition of cardiac MRI and PET images has multiple potential clinical applications, particularly in patients with coronary artery disease and cardiomyopathies. While cardiac MRI provides high spatial resolution, and precise characterization of flow and function, PET imaging adds metabolic information that can be coregistered with MRI images.

The importance of identification and quantification of the border zone of an infarct has been emphasize in recent cardiac imaging publications. The extent of border zone is a strong predictor of adverse left ventricular remodeling and lethal arrhythmias after an MI. In addition, it has been described that residual ischemia after MI is a strong predictor of adverse outcomes. However, the relationship between ischemia and border zone is not clearly understood. We have previously demonstrated the potential of chronic low dose vasodilator therapy to decrease the volume of border zone over time, a finding that suggests a potential role of combined high resolution scar and perfusion mapping in predicting response to specific treatment strategies in ischemic heart disease. In addition, combined PET MR acquisition may allow for assessment of any associations between border zone ischemia and myocardial strain, which may enhance our understanding of myocardial hybernation, and provide potential goals for treatment strategies. Compared to PET, MR has the ability to assess whether a region of ischemia and scar is transmural or not, and to map areas of core and border zone infarct. The relationship between ischemia and border zone may be an important consideration in determining whether tissue in the border zone can be salvaged. In patients with cardiac sarcoidosis and myocarditis, it is well established that abnormal cardiac MR delayed enhancement and FDG uptake are important features for diagnosis, prognosis and for guiding therapy. However, the mismatch between these abnormalities has not been interrogated. Quantification of delayed enhancement areas that do not correspond to FDG uptake could be a novel biomarker for quiescent or chronic disease, and may have important role in patient management. Another area of potential application for combined PET-MR imaging is metabolic diseases and obesity. MRI has the ability to quantify myocardial strain and vessel wall abnormalities, which can be combined with PET information on cardiac metabolism and vessel wall information to aid on characterization of obesityrelated organ damage. Combined FDG-PET acquisition with morphologic characterization of atherosclerotic plaque can also be combined with morphologic markers of inflammation, including atherosclerotic plaque

#### 10.2 Preliminary studies:

Positron emission tomography (PET) has contributed significantly to the advances in our understanding of cardiac physiology and pathophysiology for more than 20 years. In addition to being a powerful research tool in cardiology, recent technical development and improved availability facilitated also its routine clinical use in cardiology. PET is the most reliable non-invasive tool for the identification of myocardial viability and also allows accurate assessment of myocardial perfusion and coronary artery disease (CAD), which is known to be the leading cause of mortality in adults. Imaging of myocardial viability with PET has been shown to identify heart failure patients who are at increased risk of death, which can be effectively reduced by surgical treatment.

components, and contrast enhancement with ferumoxytol, a marker of vessel wall inflammation.

Magnetic resonance imaging (MRI) has rapidly developed into a versatile tool for investigating cardiovascular diseases, especially for the evaluation of cardiac structure, assessment of ventricular function, and detection of myocardial infarction. Therefore, the combination of this technique without ionizing

radiation with PET is attractive in many applications.

To perform a combined analysis of sequential MRI and PET studies, images must be aligned accurately in the spatial domain. However, a particular challenge in cardiac

studies is that the three spatial dimensions must be supplemented with a time dimension in order to correct for continuous motion during respiratory and cardiac

cycles. Cardiac gating is routine in MRI and also possible in PET. Moreover, the integration of respiratory triggering is achieved using "navigators" (MRI) or list-mode acquisitions (PET). However, variable acquisition times between PET and MRI cause additional problems for exact timing of events. MRI scans are typically performed within few seconds during breath-holds while PET scans have a

minimum duration of 5 min. However, spatial co-registration is rarely addressed in studies using separate, sequential MRI and PET scans. Misalignment is mostly caused by significant patient motion, respiration, and cardiac contraction. The first two are very challenging, as they are involuntary and can produce irregular patterns. In their review, Mäkela et al. summarized the co-registration accuracy for intra- and intermodal cardiac applications. For alignment of repeated MRI acquisitions accuracies of 1.5–3.0 mm were reported. Co-registration

accuracy of repeated PET studies was on the order of 1.0-2.5 mm. Finally, alignment of gated PET with gated MRI images showed an accuracy of  $2.0\pm1.6$  mm. In another study a misalignment of  $2.8\pm0.5$  mm was calculated using

thorax and lung surfaces. Co-registration of any data not acquired simultaneously is therefore a major problem in inter- and intra-modal examinations.

#### Assessment of heart failure

Ventricular function

Determination of LV function in gated PET studies is based on the use of partial volume effects. As the effective spatial resolution in clinical cardiac PET scans is approximately 6– 10 mm FWHM (full-width at half-maximum), changes in

wall thickness can be estimated in terms of changes in regional count rates during cardiac contraction. Using algorithm-dependent assumptions, such as homogeneous

tracer distribution over the myocardial wall, geometrical models can be used to estimate endo- and epicardial borders. This approach has been extensively implemented and validated in SPECT imaging and has also been

used in comparative MRI and PET studies. However, while being technically feasible, the accuracy of the assessment of global and regional LV function by PET

is limited by the low resolution of the PET compared to that of MRI. Here, MRI is clearly the modality-of-choice to quantitate cardiac function, such as volumes, mass, ejection fraction and regional wall thickening. Determination of LV function is essential for the diagnosis of heart failure and its prognostic value is well established. Therefore, its combination with any other imaging parameter is likely to provide incremental information.

#### Myocardial viability

Ischemic myocardium that is dysfunctional but viable has the potential for recovery of contractile function after revascularization. Evaluation of myocardial glucose utilization with 18F-FDG PET is considered as the most reliable tool to assess myocardial viability. Its quantitative nature allows assessment of the amount of viable tissue as a continuum from fully viable, through partially viable in the

areas of non-transmural infarction, to non-viable scar. Contrast-enhanced MRI appears to be a promising alternative capable of visualizing transmural distribution of viable and infarcted myocardium with excellent spatial resolution. Contrast-enhanced MRI of myocardial infarction is based on the delayed-enhancement technique using inversion-recovery prepared T1-weighted gradient-echo pulse

sequences after intravenous administration of Gd-DTPA. Infarcted myocardium appears enhanced relative to normal myocardium when imaged with a delay (typically 5–20 min) after intravenous injection of the contrast agent due to

different wash-out kinetics. A comparison of delayed-enhancement MRI with 18FFDG PET and 13NH3 in 31 patients with ischemic heart failure revealed that the location and extent of infarct scarring as delineated by delayed enhancement correlated very well with the non-viable segments from PET. The main source of difference between the methods was related to the presence of non-transmural

enhancement in regions that were viable on PET. This can be explained by the higher spatial resolution of MRI compared with nuclear imaging methods that makes delayed-enhancement suitable for the detection of small areas of subendocardial infarcts. An improved contractile performance after intervention is commonly considered as the gold standard for assessing myocardial viability,

although benefits of revascularization do not appear to be limited to improved function. In an initial study by Kim et al. in 41 patients with chronic ischaemic heart disease, dysfunctional segments with less than 25% of delayed enhancement were likely to recover after complete revascularization. In contrast, segments with more than 50% of delayed enhancement had a low probability (<10%) of

functional improvement. Comparable positive predictive values (73%) for functional recovery 6 months after revascularization were found for the lack of delayed enhancement (cut-off value less than 50% transmural scar) and the presence of preserved 18F-FDG uptake (cut-off value more than 50% of normal myocardium) as assessed by PET as the reference method to detect viable vs. nonviable myocardium. A recent meta-analysis of diagnostic studies indicated

that 18F-FDG PET has a higher sensitivity than delayed enhancement MRI (92% vs. 84%) in predicting functional recovery upon revascularization, while specificities were comparable (63%). The relatively low specificity of the techniques indicates that a substantial percentage of segments that are classified as viable by the imaging

techniques do not improve after revascularization. Although there are limited data on their combined use, adjunctive PET and MRI markers of viability, such as reduced

diastolic wall thickness, lack of contractile response to inotropic stimulation with a low dose of dobutamine, preserved epicardial rim of viable myocardium, and

preserved perfusion have been proposed to help refine the classification of dysfunctional segments as clinically viable or non-viable.

In addition to improved detection of viability, multimodal imaging approaches could contribute to the clarification of the complex pathophysiological basis underlying

the LV dysfunction in ischemic heart failure. Non-invasive detection of viable myocardium in chronic LV dysfunction associated with CAD has important clinical

implications for the treatment of patients. Although limited by the lack of large randomized clinical trials, a metaanalysis of retrospective data has indicated that such patients are also at substantial risk of death, which can be

effectively reduced by successful revascularization. Furthermore, pre-operative assessment of viability may identify patients who are at low risk of serious perioperative complications. The prognostic significance of myocardial

scars detected by delayed enhancement is currently under investigation. Among 159 patients with clinical suspicion of CAD but without a history of myocardial

infarction, the presence of even small amounts of delayed enhancement was associated with a high risk of major adverse clinical events (hazard ratio 8.29 for death, acute myocardial infarction or unstable angina pectoris, hospitalization

for heart failure, and life-threatening arrhythmias requiring defibrillation) and cardiac death (hazard ratio 10.9) during a follow-up period of 16 months [50].

It is important to emphasize that delayed-enhancement MRI is specific for either acute myocardial infarction or scar of old infarction, but not for hibernating myocardium. Plain infarct size carries well-established prognostic value

that is also expected to apply to MRI. However, in contrast,

the prognostic value of PET relies on the relative comparison of flow and glucose uptake (mismatch), which has been shown experimentally and clinically to reflect

viable, but jeopardized myocardium. Several studies have indicated that there is an association between PET "mismatch" and adverse clinical outcome [3]. There is a

need for prospective clinical trials comparing measures of infarction and either hibernation or stunning obtained with MRI and PET to obtain prognostic data to better understand whether they provide complementary clinical value.

Our research team has high level of expertise in advanced cardiac MRI and cardiac PET imaging techniques and clinical applications. Dr Ordovas has multiple prior publications on viability and functional imaging and its applications in ischemic and non-ischemic heart disease. She has a previous work on border zone response to chronic vasodilator therapy. Dr Pampaloni has studied and published cardiac PET applications for perfusion and viability, with special focus on quantitative imaging.

Dr Saloner has extensive experience with cardiac MR techniques for myocardial strain imaging, and multiple publications on the topic.

Dr Michael Hope has previous publications on aortic imaging and 4d flow MR techniques for flow characterization of patients with bicuspid aortic valve.

#### 10.3 References:

#### References

Klocke FJ, Baird MG, Lorell BH, Bateman TM, Messer JV, Berman DS, et al. ACC/AHA/ASNC guidelines for the clinical use of cardiac radionuclide imaging – executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASNC Committee to Revise the 1995 Guidelines for the Clinical Use of Cardiac Radionuclide Imaging). J Am Coll Cardiol 2003;42:1318–33.

Eisner RL, Patterson RE. Attenuation correction for stress and rest PET 82Rb myocardial perfusion images. J Nucl Med 2007; 48:1912–3.

Allman KC, Shaw LJ, Hachamovitch R, Udelson JE. Myocardial viability testing and impact of revascularization on prognosis in patients with coronary artery disease and left ventricular dysfunction: a meta-analysis. J Am Coll Cardiol 2002;39:1151–8.

Swedberg K, Cleland J, Dargie H, Drexler H, Follath F, Komajda M, et al. Guidelines for the diagnosis and treatment of chronic heart failure: executive summary (update 2005): The Task Force

for the Diagnosis and Treatment of Chronic Heart Failure of the European Society of Cardiology. Eur Heart J 2005;26:1115–40.

Martinez-Moller A, Zikic D, Botnar RM, Bundschuh RA, Howe W, Ziegler SI, et al. Dual cardiac-respiratory gated PET: implementation and results from a feasibility study. Eur J Nucl Med Mol Imaging 2007;34:1447–54.

Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, et al. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Int J Cardiovasc Imaging 2002;18:539–42.

Sinha S, Sinha U, Czernin J, Porenta G, Schelbert HR.
Noninvasive assessment of myocardial perfusion and metabolism:
feasibility of registering gated MR and PET images. AJR Am J
Roentgenol 1995;164:301–7.

Mäkela T, Clarysse P, Lötjönen J, Sipilä O, Lauerma K, Hänninen H, et al. A new method for the registration of cardiac PET and MR images using deformable model based segmentation of the main thorax structures. In: Niessen W, Viergever M, editors. Medical image computing and computer-assisted intervention – MICCAI 2001. Lecture Notes in Computer Science, vol. 2208. 4th International Conference, Utrecht, The Netherlands, October 14–17, 2001. Heidelberg: Springer; 2001. p. 557–64.

Martinez-Moller A, Souvatzoglou M, Navab N, Schwaiger M, Nekolla SG. Artifacts from misaligned CT in cardiac perfusion PET/CT studies: frequency, effects, and potential solutions. J Nucl Med 2007;48:188–93.

Gould KL, Pan T, Loghin C, Johnson NP, Guha A, Sdringola S. Frequent diagnostic errors in cardiac PET/CT due to misregistration of CT attenuation and emission PET images: adefinitive analysis of causes, consequences, and corrections. J Nucl Med 2007;48:1112–21.

Souvatzoglou M, Bengel F, Busch R, Kruschke C, Fernolendt H, Lee D, et al. Attenuation correction in cardiac PET/CT with three different CT protocols: a comparison with conventional PET. Eur J Nucl Med Mol Imaging 2007;34:1991–2000.

Bluemke DA, Achenbach S, Budoff M, Gerber TC, Gersh B, Hillis LD, et al. Noninvasive coronary artery imaging: magnetic resonance angiography and multidetector computed tomography angiography: a scientific statement from the american heart association committee on cardiovascular imaging and intervention of the council on cardiovascular radiology and intervention, and the councils on clinical cardiology and cardiovascular disease in the young. Circulation 2008;118:586–606.

Khorsand A, Graf S, Frank H, Kletter K, Sochor H, Maurer G, et al. Model-based analysis of electrocardiography-gated cardiac (18)F-FDG PET images to assess left ventricular geometry and contractile function. J Nucl Med 2003;44:1741–6.

Schaefer WM, Lipke CS, Nowak B, Kaiser HJ, Reinartz P, Buecker A, et al. Validation of QGS and 4D-MSPECT for quantification of left ventricular volumes and ejection fraction from gated 18F-FDG PET: comparison with cardiac MRI. J Nucl Med 2004;45:74–9.

Bellenger NG, Davies LC, Francis JM, Coats AJ, Pennell DJ. Reduction in sample size for studies of remodeling in heart failure by the use of cardiovascular magnetic resonance. J Cardiovasc Magn Reson 2000;2:271–8.

Schinkel AF, Poldermans D, Elhendy A, Bax JJ. Assessment of myocardial viability in patients with heart failure. J Nucl Med 2007;48:1135–46.

Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, et al. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation 1999;100:1992–2002.

Klein C, Schmal TR, Nekolla SG, Schnackenburg B, Fleck E, Nagel E. Mechanism of late gadolinium enhancement in patients with acute myocardial infarction. J Cardiovasc Magn Reson 2007;9:653–8.

Klein C, Nekolla SG, Bengel FM, Momose M, Sammer A, Haas F, et al. Assessment of myocardial viability with contrastenhanced magnetic resonance imaging: comparison with positron emission tomography. Circulation 2002;105:162–7.

Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, et al. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med 2000;343:1445–53.

Kuhl HP, Lipke CS, Krombach GA, Katoh M, Battenberg TF, Nowak B, et al. Assessment of reversible myocardial dysfunction in chronic ischaemic heart disease: comparison of contrastenhanced cardiovascular magnetic resonance and a combined positron emission tomography–single photon emission computed tomography imaging protocol. Eur Heart J 2006;27:846–53.

Gerber BL, Rochitte CE, Bluemke DA, Melin JA, Crosille P, Becker LC, et al. Relation between Gd-DTPA contrast enhancement and regional inotropic response in the periphery and center of myocardial infarction. Circulation 2001;104:998–1004.

Schmidt M, Voth E, Schneider CA, Theissen P, Wagner R, Baer FM, et al. F-18-FDG uptake is a reliable predictory of functional recovery of akinetic but viable infarct regions as defined by magnetic resonance imaging before and after revascularization. Magn Reson Imaging 2004;22:229–36.

Higuchi T, Nekolla SG, Jankaukas A, Weber AW, Huisman MC, Reder S, et al. Characterization of normal and infarcted rat myocardium using a combination of small-animal PET and clinical MRI. J Nucl Med 2007;48:288–94.

Haas F, Haehnel CJ, Picker W, Nekolla S, Martinoff S, Meisner H, et al. Preoperative positron emission tomographic viability assessment and perioperative and postoperative risk in patients with advanced ischemic heart disease. J Am Coll Cardiol 1997;30:1693–700.

Kwong RY, Chan AK, Brown KA, Chan CW, Reynolds HG, Tsang S, et al. Impact of unrecognized myocardial scar detected by cardiac magnetic resonance imaging on event-free survival in patients presenting with signs or symptoms of coronary artery disease. Circulation 2006;113:2733–43.

Muzzarelli S, Ordovas KG, Cannavale G, Naeger
D, Michaels AD, Higgins CB. Potential of Delayed Gadolinium
Enhancement Magnetic Resonance Imaing for Quantification of Reverse
Remodeling of the Peri-Infarct Zone in Patients with Ischemic Cardiomyopathy Treated
with Chronic Vasodilator Therapy: Initial Experience. J Thoracic Imaging 2011 33(6): 1440-6.

Akhtar M, Ordovás KG, Martin A, Higgins CB, Michaels AD. Effect of Chronic Sustained-Release Dipyridamole on Myocardial Blood Flow and Left Ventricular Function in Patients with Ischemic Cardiomyopathy. Congestive Heart Failure 2007, 13: 130-135.

Ordovas KG, Higgins CB. Delayed contrast enhancement on MR images of myocardium: past, present, future. <u>Radiology.</u> 2011 Nov;261(2):358-74.

Moraes GL, Higgins CB, Ordovas KG. Delayed enhancement magnetic resonance imaging in nonischemic myocardial disease. J Thorac Imaging. 2013 Mar;28(2):84-92.

Ordovás KG, Reddy GP, Higgins CB. MRI in Non-ischemic Acquired Heart Disease. JMRI 2008;27(6):1195-213.

Reddy GP, Pujadas S, Ordovás KG, Higgins CB. MR Imaging of Ischemic Heart Disease.

Magn Reson Imaging Clin N Am. 2008;16(2):201-12.

Muzzareli S, Ordovas KG, Higgins CB. Cardiovascular Magnetic Resonance Imaging for the

Assessment of Heart Failure: Focus on clinical management and prognosis. JMRI 2011; 33(2): 275-86.

Muzzareli S, Ordovas KG, Meadows A, Higgins CB. Impact of Excursion of the Interventricular Septum on Left Ventricular Systolic Function and Fibrosis after Surgical Repair of Tetralogy of Fallot. Radiology 2011; 259(2): 375-83.

Karen G. Ordovas, Marcus Carlsson, Katy E. Lease, Elyse Foster, Alison K. Meadows, Alastair J. Martin, Michael Hope, Loi Do, Charles B. Higgins, Maythem Saeed, PhD. Impaired Regional Left Ventricular

Strain After Repair of Tetralogy of Fallot. JMRI 2012; 35(1): 79-85.

Peral V, Vilacosta I, de la Pena A, San Roman JA, Fernandez C, Hernandez M, Batlle E, Carreras JL, Bethencourt A, "Thallium-201 Scintigraphy and Dobutamine Echocardiography in the Assessment of Myocardial Viability," *Rev Clin Esp.* 201: 5-15, 2001.

Hernandez-Pampaloni M, Keng FY, Kudo T, Sayre J, Schelbert HR, "Abnormal Longitudinal Base to Apex Myocardial Perfusion Gradient by Quantitative Blood Flow Measurements in Patients with Coronary Risk Factors," *Circulation* 104: 522-526, 2001.

Peral V, Vilacosta I, Fernandez C, Hernandez-Pampaloni M, San Roman JA, Battle E, Merono E, Carreras JL, Bethencourt A, "Comparison of Dobutamine Echocardiography and 201-Thallium Imaging Tomography in the Assessment of Viability Considering Positron Emission Tomography as Gold Standard," *Rev Esp Cardiol*, 54: 1394-1405, 2001.

Campisi R, Nathan L, Hernandez Pampaloni M, Schoder H, Sayre J, Chaudhuri G, Schelbert H, "Coronary Microcirculatory Function in Postmenopausal Women Following Acute and Chronic Estrogen Administration," *Circulation* 105: 425-430, 2002

Hernandez-Pampaloni M, Allada V, Fishbein MC, Schelbert HR, "Assessment of Myocardial Perfusion and Viability in Infants and Children with Suspected Coronary Abnormalities by Positron Emission Tomography: Correlation with Coronary Angiography and Histopathology," *J Am Coll Cardiol* 41: 618-626, 2002.

Hernandez-Pampaloni M, Peral V, Fernandez C, Carreras JL, Merono E, Sanchez-Harguindey L, Vilacosta I. "Biphasic Dobutamine Echocardiographic Response Predicts Improvement of Left Ventricular Dysfunction After Surgical Revascularization. Comparison with positron Emission and Rest-Redistribution Tl Tomography," *I ntl J Cardi Imaging* 19;519-528,2003.

Quinones M, Hernandez-Pampaloni M, Jimenez X, Chun Y, De La Rosa R, Modelevsky T, Castellani L, Elashoff R, Schelbert H, Hsueh WA. "Coronary V asomotion Dysfunction in Early Resistance: Normalization by Ppar-Gamma Agonists," *Annals Int Med* 140: 700-708, 2004.

M Hernandez-Pampaloni, J Bax, K Morita, D Dutka, PG Camici. "Incidence of stunned, hibernating and scarred myocardium in patients with ischemic cardiomyopathy". *Eur J Nucl & Mol Imag*, 32(3):314-321, 2005.

JO Prior, A Facta, M Hernandez-Pampaloni, TH Schindler, JW Sayre, WA Hsueh, M Quinones, HR Schelbert. "Coronary circulatory dysfunction i n insulin resistance, impaired glucose tolerance and type 2 diabetes". *Circulation*, 111;18:2291-2298, 2005.

Botvinick EH, Perini R, Bural G, Chen W, Chryssikos T, Houseni M, Hernandez-Pampaloni M, Torigian DA, Alavi A. "The aging of the heart and blood vessels: a consideration of anatomy and physiology in the era of computed tomography, magnetic resonance imaging, and positron emission tomographic imaging

methods with special consideration of atherogenesis. "Semin Nucl Med, 37:2;120-143, 2007.

Well, DS, Meier JM, Mahne A, Houseni M, Hernandez-Pampaloni M, Mong A, Mishra S, Zhuge Y, Souza A, Udupa JK, Alavi A, Torigian DA. "Detection of age-related changes in thoracic structure and function by computed tomography, magnetic resonance imaging, and positron emission tomography." Semin Nucl Med. 37:2;103-119, 2007. Brothers JA, McBride MG, Seliem MA, Marino BS, Tomlinson RS, Pampaloni MH, Gaynor JW, Spray TL, Parison, SM. Evaluation of myocardial ischemia after surgical repair of anomalous aortic origin of a coronary artery in a series of pediatric patients. J Am Coll Cardiol. 2007; 50(21):2078-82. Takalkar A, Hernandez-Pampaloni M, Cheng G, Zhuang H, Alavi A. Pediatric cardiac PET imaging. PET Clinics. 2008, Volume 3:4; 587-596. Hope MD, Meadows AK, Hope TA, Ordovás KG, Reddy GP, Alley MT, Higgins CB. Images in cardiovascular medicine. Evaluation of bicuspid aortic valve and aortic coarctation with 4D flow magnetic resonance imaging. Circulation 2008;27:117(21):2818-9. Hope MD, Hope TA, Meadows AK, Ordovás KG, Urbania TH, Alley MT, Higgins CB. Clinical Evaluation of Aortic Coarctation with 4D Flow MR Imaging. JMRI 2010; 31(3):711-18. If you have a separate bibliography, attach it to the submission with your other study documents. 11.0 Sample Size and Eligibility 11.1 Number of subjects that will be enrolled at UCSF and affiliated institutions: 60 11.2 Total number of subjects that will be enrolled at all sites (Help Text updated 9/13): 60 11.3 Estimated number of people that you will need to consent and screen here (but not necessarily enroll) to get the needed subjects: 120 11.4 Explain how and why the number of subjects was chosen (Help Text updated 9/13): This is a pilot study and we anticipate a number of 50 patients to obtain data to generate a formal sample size calculation for a larger trial. 11.5 \* Eligible age range(s): 0-6 years 7-12 years ☐ 13-17 years ✓ 18+ years

| 11.6 Inclusion criteria: | |
|---|---|
| Subjects with ischemic and non-ischemic cardiac disease referred for cardiac | PET for viability imaging. |
| 11.7 Exclusion criteria: | |
| Contraindications for MRI, including cardiac pacemaker, claustrophobia, retained metallic foreign body, cochlear implant, Aneurysm clip in the brain, pregnancy and eGFR less than 45%. | |
| 11.8 There are inclusion or exclusion criteria based on gender, race o | r ethnicity: |
| O Yes • No | |
| If <b>yes</b> , please explain the nature and rationale for the restrictions: | |
| 12.0 Drugs and Devices | |
| 12.1 * Investigational drugs or biologics will be used OR approved dr<br>under this application: | ugs or biologics will be studied |
| ⊙ Yes C No | |
| 12.2 * Investigational medical devices or in vitro diagnostics will be under this application: | ised OR approved medical devices or |
| ⊙ Yes O No | |
| 12.3 * A Non-Significant Risk (NSR) determination is being requested | for an investigational device: |
| ⊙ Yes O No | |
| 12.4 Verification of IND/IDE numbers: If the sponsor's protocol does must submit documentation from the sponsor or FDA identifying Attach this documentation in the Other Study Documents section Packet. | the IND/IDE number for this study. |
| <sup>13.0</sup> Study Drug Details | |
| 13.1 List the drugs or biologics that will be studied: | |
| 13.1 List the drugs of biologics that will be studied. | |
| View Details Drug Name FDA Approved new use of approved drug. | IND Number |
| Trade Drug<br>Gadavist<br>Name: | |
| Generic Drug Name: Yes No | |
| Investigational Drug Name: | |
| Trade Drug Name: Gadavist | |
| Generic Drug Name: Gadobutrol | |

| Investigational Drug Name: | |
|---|---|
| Identify the name of the manufacturer or source of investigational drug/biologic: | |
| Is the drug supplied at no cost? | No |
| Is the Drug FDA Approved: | Yes |
| Is this a new drug or a new use of an already approved drug | No |
| Is an IND necessary | No |
| IND Number | |
| Who holds the IND: | N/A |
| IND details: | |
| If FDA Approved and an IND is not required, Please provide a rationale for exemption: | This drug is currently used in MRI exams. |
| Are you currently using this IND in another research project? | No |
| If yes, list the IRB Number(s): | |
| Will the investigational pharmacy be dispensing? | No |
| If the source is not a FDA licensed facility, provide details regarding the purity, quality, stability and sterility of the investigational drug /biologic: | |

## 14.0 Study Device Details

List the medical devices or in vitro diagnostics to be studied or used and attach any FDA or sponsor correspondence relating to the device to the application in the Study Documents section: (Note: Device category descriptions added to the Help link December, 2014)

| View<br>Details | Device Name | | Is the Device FDA<br>Approved | IDE Number |
|---|---|---|---|---|
| Е | GE PET/MRI | | No | Yes |
| Manufact | curer/Supplier of Device | | | |
| Medicare | Category | ПА | В | |
| Where w | ill the Devices Be Stored | | | |
| Will Devi | Will Devices be supplied at no Cost | | | |
| Is this a | HUD (HDE) | No | | |
| HDE Nun | nber | | | |
| Is the De | evice FDA Approved | No | | |
| | Is this a new device or a new use of an already approved device | | | |
| Is an IDE necessary | | No | | |
| IDE Num | ber | | | |
| Who hold | ds the IDE | N/A | | |

| ta |
|----|

In the opinion of the sponsor, select the level of risk associated with this device

No Significant Risk

## 15.0 Non-Significant Risk Determination for an Investigational Device

#### 15.1 Explain why the use of the device in this study poses non-significant risk:

The PET/MRI study device is classified as non-significant risk in accordance with the definition of a significant risk device provided in 21 CFR Part 812.3(m):

It is not intended as an implant; 2) is not purported or represented to be for a use in supporting or sustaining human life; 3) is not for a use of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health; 4) and it does not otherwise present a potential for serious risk to the health, safety, or welfare of a subject (refer to additional study controls below).

Additional study controls:

For parameters besides Specific Absorption Rate (SAR), the study will comply with the non-significant risk limits described in the guidance 'Criteria for Significant Risk Investigations of Magnetic Resonance Diagnostic Devices', dated July 14, 2003. For SAR parameters, the device within the study will be tested and required to comply with the risk limits identified in IEC 60601-2-33 Ed. 3.0 Medical electrical equipment – Part 2-33: Particular requirements for the basic safety and essential performance of magnetic resonance equipment for medical diagnosis, which is a FDA Recognized Consensus standard.

Attach any supporting documentation (e.g. any reports of prior investigations) at the end of the application.

| 16.0 Other Approvals and Registrations | |
|---|---|
| 16.1 * Do any study activities take place on patient care units: | |
| O Yes • No If <b>Yes</b> , attach a letter of support for the study from the involved patient care manager(s). | |
| 16.2 * Does your protocol involve any radiation exposure to patients/subjects? The UCSF Radiatio Safety Committee requires review of your protocol if it includes administration of radiation as standard of care <u>OR</u> research exposures: | |
| O Yes O No | |
| 16.3 * This study may generate genetic data that may be broadly shared (e.g. submitted to NIH fo<br>Genome-Wide Association Studies (GWAS) in dbGaP, TCGA, etc): | r |
| O Yes O No | |
| 16.4 * This study involves administration of vaccines produced using recombinant DNA technological human subjects: | es to |
| O Yes • No | |

16.5 \* This study involves human gene transfer (NOTE: Requires NIH Recombinant DNA Advisory

| Committee (RAC) review prior to CHR approval): | |
|---|---|
| O Yes • No | |
| 16.6 This study involves other regulated materials and requires approval and/or authorization from following regulatory committees: | n the |
| ☐ Institutional Biological Safety Committee (IBC) | |
| Specify BUA #: | |
| ☐ Institutional Animal Care and Use Committee (IACUC) | |
| Specify IACUC #: | |
| Radiation Safety Committee | |
| Specify RUA #: | |
| Radioactive Drug Research Committee (RDRC) | |
| Specify RDRC #: | |
| ☐ Controlled Substances | |
| 17.0 Procedures | |
| 17.1 * Procedures/Methods (Help Text updated 9/13) For clinical research list all study procedure and treatments required for this study, including when and how often they will be performed there are no clinical procedures, describe the Methods: | |
| The subjects will undergo PET/MR for study purposes after they have finished their clinically indicated PET/CT, with no additional venipuncture to the patients. | |
| We propose to use 5D MR imaging (3D in space, in time through the cardiac cycle, and in time through the respiratory cycle) to provide improved information on the location of the signal source during PET acquisition. | |
| Dynamic and static PET data will be acquired in list mode and retrospectively rebinned according to predicted location from MR data. | |
| Accelerated MR methods (including compressed sensing) will be used to give rapid assessment of volumes over time. | |
| , | |

17.2 Interviews, questionnaires, and/or surveys will be administered or focus groups will be conducted:

| O Yes • No | |
|---|---|
| List any standard instruments used for this study: | |
| Attach any non-standard instruments at the end of the application. | |
| 17.3 Conduct of study procedures or tests off-site by non-UCSF personnel: | |
| O Yes ⊙ No | |
| If yes, explain: | |
| 17.4 Sharing of experimental research test results with subjects or their care providers: | |
| O Yes O No | |
| If yes, explain: | |
| 17.5 * Specimen collection for future research and/or specimen repository/bank administration: | |
| O Yes O No | |
| 17.6 Time commitment (per visit and in total): | |
| 1 hour in the scanner. | |
| 17.7 Locations: | |
| The cardiac MRI will take place at the China Basin radiology. | |
| 17.8 Describe the resources in place to conduct this study in a way that assures protection of the and welfare of participants: | rights |
| <ol> <li>The research team will make several efforts to keep the PHI under extreme security, including the use of a coded database, password protected computers and locked cabinets, which will all be kept inside a locked office at the Parnassus campus.</li> <li>Patients are screened for prior claustrophobic symptoms using a screening form. Earplugs are provided to all patients in order to minimize the discomfort related to the loud noise.</li> <li>Loose metal objects are not allowed in the MR room. All entrances to the scanners are clearly marked with signs warning people not to enter with any metal and by each entrance there is a mobile metal detector.</li> <li>All patients fill up a screening form for any incompatible devices and metallic foreign bodies prior to entering the MR scanner room.</li> </ol> | |
| 18.0 Alternatives | |
| 18.1 Study drug or treatment is available off-study: | |
| O Yes | |

| ○ No O Not applicable | |
|---|---|
| 18.2 * Is there a standard of care (SOC) or usual care that would be offered to prospective subject UCSF (or the study site) if they did not participate: | ts at |
| • Yes • No If yes, describe the SOC or usual care that patients would receive if they choose not to participate: If patients do not participate on the study, they will still receive the standard FDG PET-CT per clinical request. | |
| 18.3 Describe other alternatives to study participation that are available to prospective subjects: | |
| Not to participate. | |
| 19.0 Dicks and Panofits | |

#### <sup>19.0</sup> Risks and Benefits

#### 19.1 \* Risks and discomforts:

The main risks to subjects for participating in this study are related to breach of confidentiality and exposure to the MRI scanner.

No significant physical, psychological, financial, or legal harm is anticipated in case subject's confidentiality is inadvertently breached.

Risks associated with the MRI study are stratified based on probability of occurrence and listed below:

#### Common:

MR imaging may cause some discomfort, such as feelings of claustrophobia and discomfort due to loud sounds of the MR instrument during the study.

#### Uncommon/Rare:

Another potential hazard of the exam is localized heating of the body due to the radio waves employed. MR scanner and the MR probes have been designed to reduce the chance of heating.

Because the MR scanner attracts iron, there is a small possibility that an iron-containing object could accidentally fly into the magnet causing injury to the patient.

The presence of some metallic implantable devices or foreign bodies represents formal contra-indication to MR imaging and exposure to the strong magnetic field may cause malfunction or dislodgement of such devices or foreign bodies, potentially harming patients. A cardiac pacemaker is one example.

Gadolinium is considered to be very safe for most people. Side effects from gadolinium itself are very rare. These side effects are usually headache and nausea. There have been a very few people who have had allergic reactions to gadolinium. Most people with allergic reactions get hives. Patients with severe kidney disease sometimes have a bad reaction to gadolinium contrast. The condition is called nephrogenic systemic fibrosis (NSF). It can cause skin to tighten or scar and can damage internal organs. Sometimes it can be life threatening. There are no reports of NSF in patients with normal kidney function.

#### 19.2 Steps taken to minimize risks to subjects:

- 1) The research team will make several efforts to keep the PHI under extreme security, including the use of a coded database, password protected computers and locked cabinets, which will all be kept inside a locked office at the Parnassus campus.
- 2) Patients are screened for prior claustrophobic symptoms using a screening form. Earplugs are provided to all patients in order to minimize the discomfort related to the loud noise.
- 3) Loose metal objects are not allowed in the MR room. All entrances to the scanners are clearly marked with signs warning people not to enter with any metal and by each entrance there is a mobile metal detector.
- 4) All patients fill up a screening form for any incompatible devices and metallic foreign bodies prior to entering the MR scanner room.
- 5) Gadolinium: There have been a very few people who have had allergic reactions to gadolinium. Most people with allergic reactions get hives. These are usually very mild and require no treatment. Sometimes people will receive Benadryl to help relieve any itching. Subjects may experience a temporary discomfort from the needle stick, bruising, and rarely infection. Before the subject undergo an MRI requiring an

| injection of gadolinium contrast, we will review his medical record for results of a blood test to check the renal function. If the subject have not had a recent laboratory test done for that purpose, we will obtain that blood test on the day of the study, without the need for an additional puncture. Based on his medical history and the results of the test, a doctor will decide whether it is safe for you to undergo the MRI. |
|---|
| 19.3 Benefits to subjects: |
| O Yes • No If yes, describe: No direct benefit for the patients; however, future patients could benefit from the combined acquisition of PET/MRI for management of their cardiac disease. |
| 19.4 Benefits to society: |
| The combined acquisition of PET/MRI may be a reliable diagnostic and prognostic tool for patients with cardiac disease. |
| 19.5 Explain why the risks to subjects are reasonable: |
| MR imaging may cause some discomfort, such as feelings of claustrophobia and discomfort due to loud sounds of the MR instrument during the study. These discomfort and risks will be outweighed by the possibility of a reliable diagnostic and prognostic tool for patients with cardiac disease. |
| 20.0 Data and Safety Monitoring Plan |
| 20.1 Describe the plan for monitoring data and safety (Help Text updated 9/13): |
| One of the study investigators will be present during the study acquisition and will document any possible adverse reaction on a log book. Dr Ordovas and Dr Pampaloni will review the log book to confirm absence of adverse events once a week. In case of a minor adverse event, CHR will be informed within one week. In the unlikely event of a significant adverse event, CHR will be informed within 24 hours. |
| One of the study investigators will be present during the study acquisition and will document any possible adverse reaction on a log book. Dr Ordovas and Dr Pampaloni will review the log book to confirm absence of adverse events once a week. In case of a minor adverse event, CHR will be informed within one week. |
| One of the study investigators will be present during the study acquisition and will document any possible adverse reaction on a log book. Dr Ordovas and Dr Pampaloni will review the log book to confirm absence of adverse events once a week. In case of a minor adverse event, CHR will be informed within one week. In the unlikely event of a significant adverse event, CHR will be informed within 24 hours. |
| One of the study investigators will be present during the study acquisition and will document any possible adverse reaction on a log book. Dr Ordovas and Dr Pampaloni will review the log book to confirm absence of adverse events once a week. In case of a minor adverse event, CHR will be informed within one week. In the unlikely event of a significant adverse event, CHR will be informed within 24 hours. 20.2 This study requires a Data and Safety Monitoring Board: O Yes No or not sure |
| One of the study investigators will be present during the study acquisition and will document any possible adverse reaction on a log book. Dr Ordovas and Dr Pampaloni will review the log book to confirm absence of adverse events once a week. In case of a minor adverse event, CHR will be informed within one week. In the unlikely event of a significant adverse event, CHR will be informed within 24 hours. 20.2 This study requires a Data and Safety Monitoring Board: O Yes O No or not sure If yes, press SAVE and CONTINUE to move to the next section of the application. |

| ☐ Biometric identifiers | |
|---|---|
| ☐ Facial photos or other identifiable images ☐ Any other unique identifier | |
| * Required for studies conducted at the VAMC | |
| 21.5 Identifiable information might be disclosed as part of study activities: | |
| <b>⊙</b> Yes <b>○</b> No | |
| If <b>yes</b> , indicate to whom identifiable information may be disclosed: | |
| ☐ The subject's medical record | |
| ▼ The study sponsor | |
| Collaborators | |
| ▼ The US Food & Drug Administration (FDA) | |
| <ul><li>Others (specify below)</li><li>A Foreign Country or Countries (specify below)</li></ul> | |
| A Foreign Country of Countries (specify below) | |
| If <b>Others</b> , specify: | |
| 21.6 Indicate how data are kept secure and protected from improper use and disclosure (check all apply): NOTE: Whenever possible, do not store subject identifiers on laptops, PDAs, or other portable devices. If you collect subject identifiers on portable devices, you MUST encrypt the d | |
| ☐ Data are stored securely in My Research | |
| ✓ Data are coded; data key is destroyed at end of study | |
| ☑ Data are coded; data key is kept separately and securely | |
| ☑ Data are kept in a locked file cabinet<br>— | |
| ☑ Data are kept in a locked office or suite | |
| <ul><li>✓ Electronic data are protected with a password</li><li>☐ Data are stored on a secure network</li></ul> | |
| ☐ Data are collected/stored using REDCap or REDCap Survey | |
| □ Data are securely stored in OnCore | |
| 21.7 Additional measures to assure confidentiality and protect identifiers from improper use and disclosure, if any: | |
| 21.8 This study may collect information that State or Federal law requires to be reported to other or ethically requires action: | officials |
| O Yes • No | |
| Explain: | |
| 21.9 This study will be issued a Certificate of Confidentiality: | |
| O Yes ⊙ No | |
| <sup>22.0</sup> Subjects | |

| 22.1 Check all types of subjects that may be enrolled: |
|---|
| ✓ Inpatients ✓ Outpatients □ Healthy volunteers □ Staff of UCSF or affiliated institutions |
| 22.2 Additional vulnerable populations: |
| Children Subjects unable to consent for themselves Subjects unable to consent for themselves (emergency setting) Subjects with diminished capacity to consent Subjects unable to read, speak or understand English Pregnant women Fetuses Neonates Prisoners Economically or educationally disadvantaged persons Investigators' staff Students Explain why it is appropriate to include the types of subjects checked above in this particular study: Describe the additional safeguards that have been included in the study to protect the rights and welfare of these subjects and minimize coercion or undue influence: |
| 23.0 Recruitment |
| 23.1 * Methods (check all that apply): |
| Study investigators (and/or affiliated nurses or staff) recruit their own patients directly in person or by phone. |
| lacksquare Study investigators recruit their own patients by letter. Attach the letter for review. |
| <ul> <li>Study investigators send a "Dear Doctor" letter to colleagues asking for referrals of eligible patients. If interested, the patient will contact the PI or the PI may directly recruit the patients (with documented permission from the patient). Investigators may give the referring physicians a study information sheet for the patients.</li> <li>Study investigators provide their colleagues with a "Dear Patient" letter describing the study. This letter can be signed by the treating physicians and would inform the patients how to contact the study investigators. The study investigators may not have access to patient names and addresses for mailing</li> </ul> |
| Advertisements, notices, and/or media used to recruit subjects. Interested subjects initiate contact with study investigators. Attach ads, notices, or media text for review. In section below, please explain where ads will be posted. |
| · |
| Study investigators identify prospective subjects through chart review. (Study investigators request a Waiver of Authorization for recruitment purposes.) |
| $\square$ Study investigators identify prospective subjects through chart review. (Study investigators request a |
| <ul> <li>Study investigators identify prospective subjects through chart review. (Study investigators request a Waiver of Authorization for recruitment purposes.)</li> <li>Large-scale epidemiological studies and/or population-based studies: Prospective subjects are identified through a registry or medical records and contacted by someone other than their personal</li> </ul> |

| <ul> <li>Study investigators recruit potential subjects who are unknown to them through methods such as snowball sampling, direct approach, use of social networks, and random digit dialing.</li> <li>✓ Other</li> </ul> | |
|---|---|
| If <b>Other</b> , explain: | |
| Inpatients and outpatients referred for clinically indicated FGD-PET are going to be invited for participation in this study. The investigators will explain in detail the study and will provide the informed consent to the potential subject. The investigators will clarify any doubts related to the informed consent and/or the study. | |
| 23.2 * How, when, and by whom eligibility will be determined: | |
| The patients will be approached (by phone call) by one of the investigators before they arrive at the Radiology department for the clinically indicated FGD-PET. | |
| 23.3 * How, when, where and by whom potential subjects will be approached: | |
| The investigator will look for exclusion criteria of scheduled patients for FGD-PET . The patients will be approached by phone call before their scheduled appointment at the Radiology department for the clinically indicated FGD-PET. | |
| 23.4 * Protected health information (PHI) will be accessed prior to obtaining consent: | |
| ● Yes O No | |
| Waiver of Consent/Authorization for Recruitment Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. | |
| Purposes This section is required when study investigators (and/or affiliated | |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment | |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identification. | |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identified Yes | fied: |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identified. © Yes If no, a waiver of consent/authorization is NOT needed. | fied: |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identified. • Yes If no, a waiver of consent/authorization is NOT needed. 24.2 * A waiver for screening of health records to identify potential subjects poses no more than resist to privacy for participants: | fied: |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identified by Yes If no, a waiver of consent/authorization is NOT needed. 24.2 * A waiver for screening of health records to identify potential subjects poses no more than risk to privacy for participants: | fied: |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identified. © Yes If no, a waiver of consent/authorization is NOT needed. 24.2 * A waiver for screening of health records to identify potential subjects poses no more than risk to privacy for participants: © Yes If no, a waiver of authorization can NOT be granted. | fied: |
| Purposes This section is required when study investigators (and/or affiliated nurses or staff) recruit their own patients directly. 24.1 * Study personnel need to access protected health information (PHI) during the recruitment and it is not practicable to obtain informed consent until potential subjects have been identificated. ② Yes If no, a waiver of consent/authorization is NOT needed. 24.2 * A waiver for screening of health records to identify potential subjects poses no more than risk to privacy for participants: ③ Yes If no, a waiver of authorization can NOT be granted. 24.3 * Screening health records prior to obtaining consent will not adversely affect subjects' right welfare: | fied: |

| ✓ Names ✓ Dates | |
|---|---|
| Postal addresses | |
| <ul><li>✓ Phone numbers</li><li>☐ Fax numbers</li></ul> | |
| Email addresses | |
| ☐ Social Security Numbers* | |
| Medical record numbers | |
| Health plan numbers | |
| Account numbers | |
| License orcertificate numbers | |
| ☐ Vehicle ID numbers | |
| Device identifiers or serial numbers | |
| ☐ Web URLs | |
| ☐ IP address numbers | |
| ☐ Biometric identifiers | |
| Facial photos or other identifiable images | |
| Any other unique identifier | |
| □ None | |
| Note: HIPAA rules require that you collect the minimum necessary. | |
| 24.5 * Describe any health information that will be collected prior to obtaining informed consent: | |
| 24.5 Describe any health information that will be conected prior to obtaining informed consent. | |
| Name, phone number and presence of contraindications (history of cardiac pacemaker, retained metallic foreign body, cochlear implant, aneurysm clip in the brain, claustrophobia, pregnancy and eGFR less than 45%) to the MR exam. | |
| Note: HIPAA requires that you collect the minimum necessary. | |
| 24.6 * Describe your plan to destroy the identifiers at the earliest opportunity consistent with the research or provide a health or research justification for retaining the identifiers, or indicate at explain that retention is required by law: | nd |
| As soon as this study is finished, all the data will be destroyed, physically and virtually. | |
| 25.0 Informed Consent | |
| 25.1 * Methods (check all that apply): | |
| _ | |
| Signed consent will be obtained from subjects and/or parents (if subjects are minors) | |
| ☐ Verbal consent will be obtained from subjects using an information sheet or script | |
| Electronic consent will be obtained from subjects via the web or email | |
| ☐ Implied consent will be obtained via mail, the web or email | |
| ☐ Signed consent will be obtained from surrogates | |
| lacksquare Emergency waiver of consent is being requested for subjects unable to provide consent | |
| ☐ Informed consent will not be obtained | |
| 25.2 * Process for obtaining informed consent: | |

| An investigator will invite potential patients that were referred for clinically indicated FGD-PET for study participation before their exam. |
|---|
| 25.3 * How investigators will make sure subjects understand the information provided to them: |
| Investigators will talk in a lay language and will be available to clarify any doubts regarding any questions. |
| <sup>26.0</sup> Financial Considerations |
| 26.1 Subjects payment or compensation method (check all that apply): |
| Payments will be (check all that apply): Subjects will not be paid Cash Check Debit card Gift card Reimbursement for parking and other expenses Other: Specify Other: 26.2 Describe the schedule and amounts of payments, including the total subjects can receive for completing the study. If deviating from recommendations in Subject Payment Guidelines, include specific justification below. |
| Subjects will not be paid. |
| 26.3 Costs to Subjects: Will subjects or their insurance be charged for any study procedures? |
| O Yes No If <b>yes</b> , describe those costs below, and compare subjects' costs to the costs associated with alternative care off-study. Finally, explain why it is appropriate to charge those costs to the subjects. |
| 27.0 CTSI Screening Questions |
| 27.1 * This study will be carried out at one of the UCSF Clinical Research Services (CRS) centers or will utilize CRS services. CRS centers are at the following sites: SFGH Clinical Research Center Moffitt Adult Clinical Research Center Moffitt Hospital Pediatrics & NCRC Mount Zion Hospital Clinical Research Center Tenderloin Center CHORI Children's Hospital Pediatrics & Adult Clinical Research Center Kaiser Oakland Research Unit SF VA Medical Center Clinical Research Unit Please note: Effective 3/1/14, the CRS form will no longer be completed and submitted in iRIS. The CRS budget request form can be found at: https://accelerate.ucsf.edu/files/crs/BudgetRequest2015.docx. Follow the instructions on the form to submit. Even if you click 'Yes' to this question, the form will no longer proceed to the Clinical Research Services (CRS) Application Form section. |

| O Yes ⊙ No |
|------------------------------------------------------|
| 27.2 This project involves community-based research: |
| O Yes O No |
| 27.3 This project involves practice-based research: |
| O Yes • No |

## 28.0 End of Study Application

28.1 End of Study Application Form To continue working on the Study Application: Click on the section you need to edit in the left-hand menu. Remember to save through the entire Study Application after making changes. If you are done working on the Study Application: Click Save and Continue. If this is a new study, you will automatically enter the Initial Review Submission Packet form, where you can attach consent forms or other study documents. Review the Initial Review Submission Checklist for a list of required attachments. Answer all questions and attach all required documents to speed up your approval.